CLINICAL TRIAL: NCT07202676
Title: Factors Associated With the Quality of Life of Nursing Home Residents in Vietnam: A Cross-Sectional Study
Brief Title: Quality of Life (QOL), Nursing Home Residents, Vietnam.
Acronym: QOLNHVN
Status: Recruiting | Type: Observational
Sponsor: Nguyen Thi Thu Trang (Other)
Collaborators: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Sponsor-Investigator, Nguyen Thi Thu Trang, Principal Investigator, National Taipei University of Nursing and Health Sciences
Organization: National Taipei University of Nursing and Health Sciences (Other)
Other Study IDs: QOL - TRANG- 001
Record Dates: First submitted 2025-08-25; First posted 2025-10-02 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Quality of Life
Keywords: quality of life (QoL); nursing homes; activity daily living

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nursing home residents aged 60+: This cohort consists of older adults aged 60 years and above residing in selected nursing homes in Hanoi, Vietnam, who have lived in the facility for at least three months, scored within the normal range on the Montreal Cognitive Assessment (MoCA), and provided informed consent. Participants will complete structured face-to-face interviews using standardized instruments to assess quality of life, functional status, nutrition, depression, and perceived social support. No intervention will be administered, as this is an observational study.

SUMMARY:
Vietnam's rapidly aging population has increased the demand for institutional care, highlighting the importance of understanding quality of life (QoL) among older adults in nursing homes. This cross-sectional study, conducted in 2025 in Hanoi, will explore associations between QoL and factors such as demographics, health status, and social support. Data will be collected through structured interviews using validated tools (e.g., WHOQOL-BREF, Barthel Index, MSPSS, MNA-SF, NRS, GDS-15) and analyzed with descriptive and inferential statistics. The study expects to show that functional independence and strong social support are linked to better QoL. Findings will provide evidence to guide nursing practice, care planning, and policy development for older adults in Vietnam's long-term care facilities.

DETAILED DESCRIPTION:
Background: The aging of Vietnam's population has led to a growing demand for institutional care, underscoring the need to understand the quality of life (QoL) among older adults living in nursing homes. This study aims to identify and analyze factors associated with QoL, with a focus on demographic characteristics, health- related status, and perceived social support.

Methods: A cross-sectional study will be conducted in 2025 using convenience sampling from selected nursing homes in Hanoi. Participants will be aged 60 years or older, have resided in the facility for at least three months, be cognitively capable of communication, and provide informed consent. Data will be collected via structured face-to-face interviews using standardized instruments, including the WHOQOL- BREF, Barthel Index, Multidimensional Scale of Perceived Social Support (MSPSS), Mini Nutritional Assessment (MNA-SF), Numerical Raiting Scale (NRS) and Geriatric Depression Scale (GDS-15). SPSS version 27 will be used for data analysis, employing descriptive and inferential statistics such as t-tests, ANOVA, Pearson's correlation, and multiple linear regression.

Expected Results: It is anticipated that higher levels of functional independence and perceived social support will be positively associated with better QoL outcomes.

Expected Conclusion/Implications: Findings from this study are expected to contribute to evidence-based nursing practice and inform care planning and policy- making to improve the well-being of older adults in long-term care facilities in Vietnam.

ELIGIBILITY:
Inclusion Criteria:

* - Aged 60 years or older
* Had resided in a nursing home for at least 3 months
* Capable of verbal communication and able to participate in a face-to-face interview - Had adequate cognitive function to complete the questionnaire, defined as a MoCA score ≥ 26
* Provided written informed consent

Exclusion Criteria:

* Has significant language barriers, such as being unable to communicate in Vietnamese or only speaking a minority language for which the research team does not have an appropriate interpreter.
* Is experiencing acute medical conditions requiring emergency treatment or is under medical isolation as required by public health regulations (e.g., in cases of acute infectious diseases).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Other
Study Population: Older adults aged 60 and above residing in nursing homes in Hanoi in 2025. Facilities will be selected based on logistical feasibility and formal approval from the director. They provide long-term or day-care services, including assistance with ADLs, medical supervision, rehabilitation, and social activities, accommodating residents with varying physical and cognitive abilities.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Factors associated with quality of life of nursing home residents in Vietnam | 3 months after baseline
  WHOQOL-BREF (Vietnamese validated version, 26 items) is a widely used instrument for assessing quality of life across four domains: Physical Health (7 items), Psychological (6 items), Social Relationships (3 items), and Environment (8 items), along with 2 global items on overall quality of life and general health. Each item is rated on a 5-point Likert scale, and domain scores are transformed to a 0-100 scale, with higher scores indicating better quality of life. In this study, all 26 items will be administered to older adults residing in nursing homes to evaluate multidimensional quality of life, enabling analysis of its associations with demographic characteristics, health status, and perceived social support.

CONTACTS AND LOCATIONS:
Overall Officials: Lai Ting, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Bach Nien Thien Duc Nursing home, Dien Hong Nursing Home, Nhan Ai Nursing Home, Social Protection Center Hanoi 1, Social Protection Center Hanoi 2, Social Protection Center Hanoi 3, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the sensitive nature of personal health and social information collected from older adults in nursing homes. Data will be kept confidential and used solely for the purposes of this study.

DOCUMENTS (1):
  • Informed Consent Form (2025-09-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT07202676/ICF_000.pdf